CLINICAL TRIAL: NCT03067324
Title: Quality Control of Pancreatic Islet Intended to Islet Graft
Brief Title: Quality Control of Pancreatic Islet Intended to Islet Graft Cells Intended to Stabilot Islet Graft Protocol
Acronym: ISLET CHIP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC14.041
Record Dates: First submitted 2017-02-21; First posted 2017-03-01 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Pancreatic Islet Quality Control
Keywords: Islet Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — pancreatic islet cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Islet quality control after pancreatic islets isolation process is insufficient. The Islet Chip study proposes to develop a bio-sensor that will allow a multi-parametric analysis of islet graft based on measurement of islet membrane electric potential.

DETAILED DESCRIPTION:
Islet quality control after pancreatic islets isolation process is insufficient. The Islet Chip study proposes to develop a bio-sensor that will allow a multi-parametric analysis of islet graft based on measurement of islet membrane electric potential.

The project aims to :

* develop the bio-sensor necessary to measure islet membrane electric potential
* develop interface between bio-sensor and user
* correlate analysis data collected by bio-sensor with metabolic results of islet graft

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in STABILOT Pancreatic Islet cell graft protocol and willing to participate to ISLET CHIP

Exclusion Criteria:

* Patients not enrolled in STABILOT Pancreatic Islet cell graft or patients that signed the form expressing their refuse to participate to ISLET CHIP.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients enrolled in STABILOT Pancreatic Islet cell graft protocol and willing to participate to ISLET CHIP
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-01-11 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Beta-score | 6 months in average before second islet graft
  Beta-score in continuous variable, using the last Beta-score known before the second islet graft. Beta-score is a composite score that reflects pancreatic islet graft function after transplantation and measured from the following criteria: severe hypoglycemia, HbA1c, stimulated C-peptide, fasting glucose, insulin dose or oral diabetes, glycemic variability.

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine LABLANCHE, MD, PhD, Principal Investigator — University Hospital, Grenoble; Bogdan CATARGI, MD, PhD, Study Director — University Hospital, Bordeaux
Locations (8):
- France (7):
  - Besançon University Hospital, Besançon
  - Clermont Ferrand University hospital, Clermont-Ferrand
  - Grenoble University Hospital, Grenoble
  - Lyon University Hospital, Lyon
  - Montpellier University Hospital, Montpellier
  - Nancy University hospital, Nancy
  - University hospital of Strasbourg, Strasbourg
- Geneva University Hospital, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kusnik-Joinville O, Weill A, Salanave B, Ricordeau P, Allemand H. Prevalence and treatment of diabetes in France: trends between 2000 and 2005. Diabetes Metab. 2008 Jun;34(3):266-72. doi: 10.1016/j.diabet.2008.01.005. Epub 2008 Jun 3. PMID 18524662
- [Background] Gruessner RW, Gruessner AC. The current state of pancreas transplantation. Nat Rev Endocrinol. 2013 Sep;9(9):555-62. doi: 10.1038/nrendo.2013.138. Epub 2013 Jul 30. PMID 23897173
- [Background] Ricordi C, Lacy PE, Finke EH, Olack BJ, Scharp DW. Automated method for isolation of human pancreatic islets. Diabetes. 1988 Apr;37(4):413-20. doi: 10.2337/diab.37.4.413. PMID 3288530
- [Background] Lablanche S, Borot S, Wojtusciszyn A, Bayle F, Tetaz R, Badet L, Thivolet C, Morelon E, Frimat L, Penfornis A, Kessler L, Brault C, Colin C, Tauveron I, Bosco D, Berney T, Benhamou PY; GRAGIL Network. Five-Year Metabolic, Functional, and Safety Results of Patients With Type 1 Diabetes Transplanted With Allogenic Islets Within the Swiss-French GRAGIL Network. Diabetes Care. 2015 Sep;38(9):1714-22. doi: 10.2337/dc15-0094. Epub 2015 Jun 11. PMID 26068866
- [Background] Lebreton F, Pirog A, Belouah I, Bosco D, Berney T, Meda P, Bornat Y, Catargi B, Renaud S, Raoux M, Lang J. Slow potentials encode intercellular coupling and insulin demand in pancreatic beta cells. Diabetologia. 2015 Jun;58(6):1291-9. doi: 10.1007/s00125-015-3558-z. Epub 2015 Mar 19. PMID 25788295
- [Background] Renaud S, Catargi B, Lang J. Biosensors in diabetes : how to get the most out of evolution and transpose it into a signal. IEEE Pulse. 2014 May-Jun;5(3):30-4. doi: 10.1109/MPUL.2014.2309577. PMID 24838208